CLINICAL TRIAL: NCT00152425
Title: A Phase III Multi-national, Multi-centre, Double-blind Placebo-controlled Parallel Group, 26 Week Study to Assess the Maintenance of Clinical Response to Humanised Anti-TNF PEG Conjugate, CDP870 400 mg sc, (Dosed 4-weekly From Weeks 8 to 24), in the Treatment of Patients With Active Crohn's Disease Who Have Responded to Open Induction Therapy (Dosed at Weeks 0, 2 and 4) With CDP870
Brief Title: Study to Test the Effect of CDP870 in the Treatment of Crohn's Disease Over 26 Weeks, Comparing CDP870 to a Dummy Drug (Placebo), Following 3 Doses of Active Drug (CDP870).
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: C87032
Record Dates: First submitted 2005-09-07; First posted 2005-09-09 (Estimated); Last update posted 2013-09-09 (Estimated); Status verified 2010-07

CONDITIONS: Crohn's Disease
Keywords: Crohn's disease, CDP870, CDAI, clinical response, remission, Certolizumab Pegol, Cimzia
MeSH Terms: conditions — Crohn Disease; Anemia, Dyserythropoietic, Congenital | interventions — Certolizumab Pegol

INTERVENTIONS:
Drug: Certolizumab Pegol (CDP870)

SUMMARY:
A 26 week maintenance study of CDP870 in Crohn's disease

ELIGIBILITY:
Inclusion Criteria:

* Definitive diagnosis of Crohn's disease confirmed (at least 3 months prior to study entry) either by radiological, endoscopic or histological evidence, affecting the terminal ileum (L1), colon (L2) or ileocolon (L3)*. * Vienna Classification (1998)
* Active Crohn's disease (≥ 220 and ≤ 450) scored over the 7 days prior to the first dose of study drug.
* Patients aged 18 years or above at screening.

Exclusion Criteria:

* Crohn's Disease Related
* Fistula abscess present at screening.
* Stricturing type disease with symptoms or signs of non-inflammatory mechanical obstruction or bowel perforation in last 3 months.
* Short bowel syndrome.
* Functional colostomy or ileostomy (note: patients who have had a temporary stoma in the past, which has been reversed, are eligible to enter the study).
* Positive stool laboratory results for enteric pathogens.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 392
Dates: Start 2004-02; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Clinical response at Week 26, in the strata defined by CRP ≥ 10 mg/L.

SECONDARY OUTCOMES:
In population with CRP ≥ 10 mg/L at baseline; Time to disease progression up to and including Week 26; Proportion of patients with clinical remission at Week 26; Proportion of patients with IBDQ response at Week 26; F-36 sub-scores and change from basel

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — UCB Pharma

REFERENCES:
- [Result] Schreiber S, Khaliq-Kareemi M, Lawrance IC, Thomsen OO, Hanauer SB, McColm J, Bloomfield R, Sandborn WJ; PRECISE 2 Study Investigators. Maintenance therapy with certolizumab pegol for Crohn's disease. N Engl J Med. 2007 Jul 19;357(3):239-50. doi: 10.1056/NEJMoa062897. PMID 17634459
- [Result] Feagan BG, Reilly MC, Gerlier L, Brabant Y, Brown M, Schreiber S. Clinical trial: the effects of certolizumab pegol therapy on work productivity in patients with moderate-to-severe Crohn's disease in the PRECiSE 2 study. Aliment Pharmacol Ther. 2010 Jun;31(12):1276-85. doi: 10.1111/j.1365-2036.2010.04303.x. Epub 2010 Mar 18. PMID 20298497
- [Result] Lichtenstein GR, Thomsen OO, Schreiber S, Lawrance IC, Hanauer SB, Bloomfield R, Sandborn WJ; Precise 3 Study Investigators. Continuous therapy with certolizumab pegol maintains remission of patients with Crohn's disease for up to 18 months. Clin Gastroenterol Hepatol. 2010 Jul;8(7):600-9. doi: 10.1016/j.cgh.2010.01.014. Epub 2010 Feb 1. PMID 20117244
- [Result] Hanauer SB, Panes J, Colombel JF, Bloomfield R, Schreiber S, Sandborn WJ. Clinical trial: impact of prior infliximab therapy on the clinical response to certolizumab pegol maintenance therapy for Crohn's disease. Aliment Pharmacol Ther. 2010 Aug;32(3):384-93. doi: 10.1111/j.1365-2036.2010.04360.x. Epub 2010 May 18. PMID 20491747
- [Result] Feagan BG, Coteur G, Tan S, Keininger DL, Schreiber S. Clinically meaningful improvement in health-related quality of life in a randomized controlled trial of certolizumab pegol maintenance therapy for Crohn's disease. Am J Gastroenterol. 2009 Aug;104(8):1976-83. doi: 10.1038/ajg.2009.199. Epub 2009 May 26. PMID 19471252
- [Result] Coteur G, Feagan B, Keininger DL, Kosinski M. Evaluation of the meaningfulness of health-related quality of life improvements as assessed by the SF-36 and the EQ-5D VAS in patients with active Crohn's disease. Aliment Pharmacol Ther. 2009 May 1;29(9):1032-41. doi: 10.1111/j.1365-2036.2009.03966.x. PMID 19222413
- [Result] Feagan BG, Hanauer SB, Coteur G, Schreiber S. Evaluation of a daily practice composite score for the assessment of Crohn's disease: the treatment impact of certolizumab pegol. Aliment Pharmacol Ther. 2011 May;33(10):1143-51. doi: 10.1111/j.1365-2036.2011.04636.x. Epub 2011 Mar 28. PMID 21443536
- [Derived] Schreiber S, Lawrance IC, Thomsen OO, Hanauer SB, Bloomfield R, Sandborn WJ. Randomised clinical trial: certolizumab pegol for fistulas in Crohn's disease - subgroup results from a placebo-controlled study. Aliment Pharmacol Ther. 2011 Jan;33(2):185-93. doi: 10.1111/j.1365-2036.2010.04509.x. Epub 2010 Nov 17. PMID 21083671
- [Derived] Lewis JD. Anti-TNF antibodies for Crohn's disease--in pursuit of the perfect clinical trial. N Engl J Med. 2007 Jul 19;357(3):296-8. doi: 10.1056/NEJMe078111. No abstract available. PMID 17634466